CLINICAL TRIAL: NCT06880250
Title: Open-label Comparative Cohort Non-interventional Epidemiological Study of the Efficacy and Safety of Enzyme Replacement Therapy in Russian Patients With Fabry Disease
Brief Title: Efficacy and Safety of Enzyme Replacement Therapy in Patients With Fabry Disease
Acronym: FAVORIT
Status: Enrolling by invitation | Type: Observational
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Other Study IDs: FAVORIT
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-05

CONDITIONS: Fabry Disease
Keywords: Fabry; ERT; enzyme replacement therapy
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fabagal: Patients taking Fabagal® as the enzyme replacement therapy
- Fabrazyme: Patients taking Fabrazyme® as the enzyme replacement therapy
- Replagal: Patients taking Replagal® as the enzyme replacement therapy

SUMMARY:
The goal of this observational study is to learn how enzyme replacement therapy works in patients with Fabry disease. The main question it aims to answer is:

What medical problems do participants have?

Participants already on enzyme replacement therapy as part of their regular medical care for Fabry disease will be observed as usual. Their data will be collected by their doctor.

DETAILED DESCRIPTION:
All patients on enzyme replacement therapy could be enrolled in the study. Three medicines are currently available in Russia (Fabagal®, Fabrazyme®, Replagal®) so the patients form three cohorts.

For all patients retrospective data are collected for 12 months prior enrollment.

All patients are observed prospectively for 6 months. At the point of 6 months patients taking Fabrazyme or Replagal at the moment finish the study.

Patients on Fabagal are observed for 12 more months (up to 18 months after enrollment).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a confirmed diagnosis of Fabry disease;
* Prescribed course of enzyme replacement therapy with any drug (Fabagal, Fabrazyme, Replagal);
* Age 8 - 65 years;
* Signed informed consent of the patient and/or patient's legal representative for participation in the study and processing of personal data.

Exclusion Criteria:

* Renal replacement therapy or kidney transplantation;
* Critical illness unrelated to Fabry disease;
* Pregnancy or breastfeeding;
* Refusal of the patient (or patient's legal representative) from further participation in the study or medical care.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Russian patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Lyso-Gb3 Level | From 12 months before enrollment up to 6 months (for Fabrazyme and Replagal cohorts) or up to 18 months (for Fabagal cohort) of observation
  Level of globotriaosylsphingosine (lyso-Gb3) is measured in dried blood spots.

SECONDARY OUTCOMES:
Change from Baseline in α-GAL Activity | From 12 months before enrollment up to 6 months (for Fabrazyme and Replagal cohorts) or up to 18 months (for Fabagal cohort) of observation
  Level of α-Galactosidase (α-GAL) activity is measured in dried blood spots.
Change from Baseline in GFR | From 12 months before enrollment up to 6 months (for Fabrazyme and Replagal cohorts) or up to 18 months (for Fabagal cohort) of observation
  Glomerular filtration rate (GFR) is measured by methods available in routine medical use.
Change from Baseline in Neuropathic Pain Level | From enrollment up to 6 months (for Fabrazyme and Replagal cohorts) or up to 18 months (for Fabagal cohort) of observation
  Neuropathic pain is assessed according to verbal scale: no pain, mild pain, moderate pain, severe pain, very severe pain, intolerable pain. Corresponding value of 0, 2, 4, 6, 8, 10 is assigned.
Incidence Rate of Significant Clinical Outcomes | From enrollment up to 6 months (for Fabrazyme and Replagal cohorts) or up to 18 months (for Fabagal cohort) of observation
  Significant clinical outcomes include cardiac rhythm disturbances (atrial fibrillation, persistent supraventricular or ventricular tachycardia), heart failure, stroke, initiation of renal replacement therapy and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Moiseev, MD, Study Chair — Sechenov First Moscow State Medical University (Sechenov University)
Locations (23):
- Russia (23):
  - #13, Astrakhan
  - #27, Barnaul
  - #7, Borovichi
  - #6, Chelyabinsk
  - #21, Grozny
  - #16, Gubkin
  - #26, Irkutsk
  - #12, Ivanovo
  - #19, Kaa-Khem
  - #10, Krasnodar
  - #18, Kurgan
  - #17, Omsk
  - #15, Orenburg
  - #9, Perm
  - #23, Polevskoy
  - #2, Rostov-on-Don
  - #4, Rostov-on-Don
  - #24, Ryazan
  - #8, Saint Petersburg
  - #3, Simferopol
  - #22, Stavropol
  - #11, Ufa
  - #5, Voronezh

IPD SHARING:
Plan to Share IPD: Undecided